CLINICAL TRIAL: NCT04419909
Title: Retreatment With CTL019/CTL119 in Patients With Late Relapse of B-Cell Lymphomas
Brief Title: Retreatment With CTL019/CTL119
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 40419; 834286 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma, B-Cell
Keywords: CTL019; CTL119; CAR T-cell; CART
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Retreatment with CTL019/CTL119 (Experimental): All subjects will receive retreatment with CTL019/CTL119 and be followed per the schedule of procedures.
  Interventions: Drug: CD19 redirected autologous T cells (CTL019 or CTL119 cells)

INTERVENTIONS:
Drug: CD19 redirected autologous T cells (CTL019 or CTL119 cells) — Retreatment with CD19-directed Chimeric Antigen Receptor-modified T Cells (CART19 cells) or huCD19-directed Chimeric Antigen Receptor-modified T Cells (huCART19 cells) in subjects with late relapse of B-cell lymphomas.

SUMMARY:
This research study is designed to evaluate the effects of retreatment with CTL019/CTL119 in patients with late relapse of B-cell lymphomas.

DETAILED DESCRIPTION:
This is a single arm open label trial that will assess the safety and efficacy of retreatment with CTL019/CTL119 chimeric antigen receptor (CAR) modified T cells in patients who have late relapse of diffuse large B-cell or follicular lymphoma after achieving complete remission from prior CTL019/CTL119 treatment. Patients eligible for this protocol will have been treated initially with CTL019/CTL119 under UPCC13413/NCT02030834, have experienced a durable complete response (defined as ≥ 6 months duration), and have a residual manufactured CTL019/CTL119 product available. This protocol will serve subjects with no available potentially curative treatment options (such as autologous or allogeneic stem cell transplantation) who have a limited prognosis (months to < 2 year expected survival) with available therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Diffuse Large B-Cell Lymphoma or Follicular lymphoma, previously identified as CD19+
2. Previously treated on UPCC13413/ NCT02030834 with CTL019/CTL119, with historical manufactured product available at Penn for reinfusion
3. Previous complete response to CAR T-cells with a duration ≥ 6 months (defined as 168 days)
4. No available curative treatment options (such as autologous or allogeneic HSCT) with limited prognosis (several months to < 2 year survival) with currently available therapies.
5. Age ≥18 years
6. Creatinine < 1.6 mg/dL
7. ALT/AST < 3x upper limit of normal
8. Bilirubin < 2.0 mg/dL, unless subject has Gilbert's Syndrome (≤3.0 mg/dL)
9. Measurable or assessable disease according to the "Revised Response Criteria for Malignant Lymphoma" (Cheson et al., J. Clin. Onc., 2007)88. Patients in complete remission with no evidence of disease are not eligible.
10. Performance status (ECOG) 0 or 1.
11. Left Ventricle Ejection Fraction (LVEF) > 40% confirmed by ECHO/MUGA
12. Agree to contraceptive requirements outlined in Section 4.3.
13. Provide written informed consent.

Exclusion Criteria:

1. Uncontrolled active infection.
2. Active hepatitis B or hepatitis C infection.
3. Any uncontrolled active medical disorder that would preclude participation as outlined.
4. Class III/IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 1).
5. HIV infection.
6. Patients with active CNS involvement by malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment
7. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | At time of consent through 1 year after the subject received CTL019/CTL119
  Safety of retreatment with CTL019/CTL119 as measured by treatment-related events

SECONDARY OUTCOMES:
Overall response rate using Cheson 2007 criteria | Month 3 post-infusion
  Efficacy of retreatment with CTL019/CTL119 as measured by ORR by Cheson 2007 definitions at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Schuster, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No